CLINICAL TRIAL: NCT05536674
Title: Design, Test and Evaluate Behavioural Insights Interventions to Strengthen Demand for Immunisation in Georgia
Brief Title: SMS Reminders to Strengthen Demand for HPV Vaccination in Georgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Behavioural Insights Team (Other)
Collaborators: UNICEF (Other); National Center for Disease Control and Public Health, Georgia (Unknown); Information Technology Agency, Georgia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNICEF Georgia 2020021
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: HPV, Human Papillomavirus Viruses, Human Papilloma Virus Vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No SMS reminder (No Intervention): This group will receive no reminder
- Short SMS with no additional information (Experimental): Caregivers of girls eligible to receive the HPV vaccination in this group will receive an SMS reminder that states: "As per national immunization calendar your daughter is due her free human papilloma virus vaccine, which will protect her against cervical cancer. Contact your family doctor today to arrange an appointment."
  Interventions: Behavioral: SMS reminder for the HPV vaccination
- Short SMS + NCDC link (Experimental): Caregivers of girls eligible to receive the HPV vaccination in this group will receive an SMS reminder that states: "As per national immunization calendar your daughter is due her free human papilloma virus vaccine, which will protect her against cervical cancer. Contact your family doctor today to arrange an appointment. More information on the official NCDC website"
  Interventions: Behavioral: SMS reminder for the HPV vaccination
- SMS with "reserved for her" framing + NCDC link (Experimental): Caregivers of girls eligible to receive the HPV vaccination in this group will receive an SMS reminder that states: "As per national immunization calendar your daughter is due her free human papilloma virus vaccine, which will protect her against cervical cancer. Her vaccine is reserved at the policlinic. Contact your family doctor today to arrange an appointment. More information on the official NCDC website"
  Interventions: Behavioral: SMS reminder for the HPV vaccination
- SMS with safety information + NCDC link (Experimental): Caregivers of girls eligible to receive the HPV vaccination in this group will receive an SMS reminder that states: "As per national immunization calendar your daughter is due her free human papilloma virus vaccine, which will protect her against cervical cancer. The vaccine has been given safely to more than 118 million girls worldwide. Contact your family doctor today to arrange an appointment. More information on the official NCDC website"
  Interventions: Behavioral: SMS reminder for the HPV vaccination

INTERVENTIONS:
Behavioral: SMS reminder for the HPV vaccination — A BI-informed SMS reminder to remind caregivers of girls between 10-12 years that their daughter is due the first dose of her HPV vaccination and share information about the vaccine.
  Arms: SMS with "reserved for her" framing + NCDC link; SMS with safety information + NCDC link; Short SMS + NCDC link; Short SMS with no additional information

SUMMARY:
It is possible that achieving adequate HPV vaccination coverage will allow cervical cancer to be virtually eliminated. This is a priority for Georgia, where the burden of mortality and morbidity from cervical cancer is high and the yearly prevalence of cervical cancer is 14.5 per 100,000 population.

The objective of the intervention evaluated is to increase the uptake of the 1st dose of the HPV vaccination in Georgia. The intervention aims to achieve this by providing a SMS reminder informed by behavioural insights (BI) to remind caregivers of girls between 10-12 years that their daughter is due the first dose of her HPV vaccination, share information about the vaccine, and encourage them to book an appointment to receive the vaccination. Four different SMS messages will be compared to no SMS message.

The evaluation will be a 5-arm randomised controlled trial (RCT) which aims to answer the research question: Does each of the designed BI-informed SMS reminders increase the uptake of the first dose of the HPV vaccination among eligible girls in Georgia, compared to no reminder? Our hypothesis is that SMS reminders will increase the uptake of HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Girls
* Aged 10-12 years
* Not yet received any doses of the HPV vaccine
* With a caregiver's mobile phone number in the e-health system.

Exclusion Criteria:

* Boys
* Girls aged less than 10 or more than 12 years
* Girls with no caregiver phone number in the e-health system
* Girls who have received 1 or 2 doses of the HPV vaccine

Ages: 10 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55176 (Estimated)
Dates: Start 2022-09-13 (Estimated); Primary Completion 2022-11-12 (Estimated); Study Completion 2022-11-12 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination status | At 60 days after receiving the SMS reminder
  1st dose HPV vaccination status of the caregiver's daughter

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Behrendt, Study Director — Behavioural Insights Team

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared from the e-health modules of the National Center for Disease Control and Public Health of Georgia and Information Technology Agency. All data shared will be anonymised for analysis and aggregated for reporting, there is no risk of participant identification. Data will include HPV vaccination status, the version of the SMS reminder received, and age. The data will not include information on patients' names, addresses, location, ethnicity, phone numbers, or any information on medical conditions.

REFERENCES:
- [Derived] Daly N, Merriam S, Tagliaferri G, Tomsa S, Bianco VM, Gamgebeli L, Lortkipanidze N. Effectiveness of SMS reminders to increase demand for HPV immunisation: a randomised controlled trial in Georgia. BMJ Open. 2025 Nov 13;15(11):e087080. doi: 10.1136/bmjopen-2024-087080. PMID 41248345